CLINICAL TRIAL: NCT03052998
Title: Ivermectin Treatment in Patients With Onchocerciasis-associated Epilepsy: A Randomized Clinical Trial
Brief Title: Ivermectin Treatment in Patients With Onchocerciasis-associated Epilepsy
Acronym: OAETREAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Robert Colebunders (Other)
Responsible Party: Sponsor-Investigator, Robert Colebunders, Professor infectious diseases, Universiteit Antwerpen
Organization: Universiteit Antwerpen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B300201730821; ERC grant No.671055 (Other Grant/Funding Number: European Research Council)
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Ivermectin; Onchocerciasis; Epilepsy
MeSH Terms: conditions — Onchocerciasis; Epilepsy | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivermectin (Active Comparator): Ivermectin and anti-epileptic treatment
  Interventions: Drug: Ivermectin
- no treatment (No Intervention): only anti-epileptic treatment

INTERVENTIONS:
Drug: Ivermectin — Effect of Ivermectin on frequency of seizures
  Other Names: anti-epileptic drugs
  Arms: Ivermectin

SUMMARY:
Many studies have reported an association between epilepsy, including Nodding Syndrome (NS), and onchocerciasis (river blindness). A high prevalence of epilepsy has been noted particularly in onchocerciasis hyperendemic areas where onchocerciasis is not or insufficiently controlled with mass Ivermectin distribution. There is evidence that increasing the coverage of Ivermectin reduces the incidence of epilepsy and anecdotal evidence suggests a reduction in seizure frequency in onchocerciasis associated epilepsy (OAE) patients who receive Ivermectin. Finding an alternative treatment for epilepsy in these patients will have major consequences.

Objective

To assess whether Ivermectin treatment decreases the frequency of seizures and leads to seizure freedom in OAE patients, including patients with NS. If we are able to demonstrate such an effect this would be an extra argument that Onchocerciasis is causing epilepsy and that therefore we should increase our efforts to eliminate onchocerciasis.

Methods

We will conduct a randomized clinical trial in the Democratic Republic of Congo (DRC) to compare seizure freedom in onchocerciasis infested epilepsy patients who receive immediate Ivermectin treatment with delayed (after four months) Ivermectin treatment. All participants will simultaneously receive anti-epileptic drugs (AEDs) according to local guidelines for epilepsy treatment. The primary endpoint is seizure freedom defined as no seizures during the fourth month of follow-up. Secondary endpoint is significant (>50%) seizure reduction compared to baseline seizure frequency. Reduction of seizures will be compared between Ivermectin and non-Ivermectin arms.

Current status

Start of enrolment is planned from March 2017 and we expect to have enrolled all 110 participants by August 2017. Results are expected early 2018.

Discussion

If Ivermectin treatment, in addition to AEDs, is able to lead to seizure freedom or significantly reduces seizure frequency in OAE patients this will have major consequences for epilepsy treatment in Onchocerciasis endemic regions. Ivermectin is donated for free, and in non Loa-Loa endemic regions has negligible side effects. Reducing the burden of epilepsy will have a major impact on quality of life and socio-economic status of families with affected members in Africa.

DETAILED DESCRIPTION:
Introduction

Many studies have reported an association between epilepsy, including nodding syndrome (NS), and onchocerciasis. A meta-analysis of African population-based surveys showed a variation in epilepsy prevalence consistent with onchocerciasis prevalence, with epilepsy prevalence being increased, on average, by 0.4% for each 10% increase in onchocerciasis prevalence. NS is an epileptic disorder occurring in children in onchocerciasis (river blindness) endemic regions, initially only observed in South Sudan, Uganda and Tanzania. NS occurs in previously health children, aged mainly between 5-18 years and is characterized by head-nodding, an atonic epileptic seizure. Individuals may also develop other types of seizures and stunted growth. NS should be considered part of a spectrum of onchocerciasis associated epileptic (OAE) disorders. We recently suggested that these epileptic disorders share etiological factors related to Onchocerca volvulus (OV) infection and therefore considered Ivermectin, used to treat Onchocerciasis, as a treatment option for OAE.

One dose of Ivermectin eliminates microfilariae very rapidly. A mathematical model predicted that microfilariaedermia would be reduced by half 24 h after the intake of Ivermectin. Therefore, if the microfilariae load plays an important role in causing OAE, it may be that Ivermectin also has a rapid effect on the frequency of seizures.

Ivermectin treatment may decrease seizure frequency in patients with OAE In a study in Kabarole district in Uganda in 1992, 34/91 (37%) patients reported some decrease in either the frequency or severity of seizures after one dose of Ivermectin (150 µg/kg). After being treated with Ivermectin, 13 (14%) individuals had no seizures for 3.7 months (on average). Seizures were unchanged in 51 (56%), and worsened in 6 (7%). In a recent trial in the DRC, comparing Moxidectin (an anti-OV experimental drug with a longer half-life than Ivermectin) with Ivermectin, 6 (80%) out of 7 OV infested patients with epilepsy became seizure free after treatment with Moxidectin or Ivermectin (the randomization code has not been broken yet). In one person seizure frequency was significantly reduced over the 18 month follow-up period. In this person, microfilariae remained present in skin snips, though at a lower level than before the onchocerciasis treatment. In all subjects who became seizure free, the skin snips too became microfilaria free.

To assess whether Ivermectin treatment may reduce the frequency of seizures and leads to seizure freedom, we intend to conduct a short proof of concept randomized clinical trial to compare immediate Ivermectin treatment with delayed (after 4 months) Ivermectin treatment in onchocerciasis infested persons with epilepsy. The primary outcome is seizure freedom at 4 months. Reducing the burden of epilepsy will have a major impact on quality of life and socio-economic status of families with affected members in Africa. If we are able to demonstrate an effect of Ivermectin on the frequency of seizures, this would be an extra argument that Onchocerciasis is causing epilepsy and that therefore we should increase our efforts to eliminate onchocerciasis.

Methods

Study design

This is a proof of concept randomized treatment trial consisting of 2 treatment arms, immediate (arm A) and delayed (4 months later) Ivermectin treatment (arm B). A computer-based, pre-planned age and frequency of seizures stratified randomization list will be used. The trial will not be placebo-controlled as this will be costly and we do not expect this to greatly influence reporting of seizures, our primary outcome. Epilepsy patients in both arms will additionally receive anti-epileptic drugs (AED) following local guidelines of epilepsy treatment in DRC. Study investigators collecting and analysing data will be blinded for treatment.

Study population, setting and enrollment.

The trial will take place in selected villages in the Logo health zone an onchocerciasis endemic region in the Ituri province in the DRC in areas were so far mass Ivermectin administration has not been implemented but where the National onchocerciasis program is planning to start community directed distribution of Ivermectin in 2017. Pilot studies by our group in this area show prevalence estimates of OAE of approximately 5%.

Before starting, the village chief and community health workers will be informed on the purpose and specifics of our study. When permission is obtained our medical team will visit the village and set up a mobile clinic. Patients that may fulfil eligibility criteria are selected and examined for a screening visit after informed consent is obtained from patient and/or caretaker in the local language (Alur). If the patient fulfils enrolment criteria he/she is invited to participate in the treatment trial. Detailed information about the trial is given in local language and enrollment informed consent is obtained.

The study population consists of epilepsy patients of 5 years and above with onchocerciasis and without other obvious risk factors for epilepsy.

Screening of epilepsy patients for OV infection

After informed consent is obtained , trial candidates with epilepsy will be tested for the presence of antibodies to the parasite antigen Ov16 with the Onchocerciasis IgG4 rapid test (SD BIOLINE Onchocerciasis IgG4 rapid test, Alere, Standard Diagnostics, Inc.; Yongin, Republic of Korea). Moreover, a skin snip will be taken from the left and right iliac crests with a Holtz corneoscleral punch (2mm). One sterilized punch will be used per subject. Each snip will be weighed on an analytical balance and incubated for 24 hours in isotonic saline in a well of a flat-bottomed microtitre plate. The microfilariae that emerged will be counted using an inverted microscope. The number of microfilaria in each well and the weight of the associated skin snip before incubation will be recorded. The mean of the skin microfilarial (mf) density = mf count/weight of snip across all 4 skin snips will be calculated and recorded as mf/mg. Skin biopsies will further be stored in 90% ethanol to be tested for Ov by an in-house PCR method.

Diagnosis of Onchocerciasis infection will be made when microfilaria are detected in skin snip and/or antibodies to the parasite antigen Ov16 are detected.

To identify eligible epilepsy patients with generalized tonic clonic seizures we will use a 10-item Epilepsy Questionnaire previously used in international epilepsy prevalence studies. A persons identified on the basis of this questionnaire as possibly a person with epilepsy will be examined by a neurologist to make an accurate diagnosis according to definitions proposed by the International League Against Epilepsy (ILAE). A case of epilepsy will be defined as a patient who had (1) at least two times, unprovoked and without fever, lost consciousness with convulsions with a minimal time difference of 24h between the two events or (2) one unprovoked seizure and a probability of future seizures similar to the general recurrence risk after 2 unprovoked seizures. Detailed questions among others on the age of seizure onset, seizure frequency, family history of seizures are part of the baseline questionnaire.

Blood samples will be tested for Taenia solium antibodies and antigen, but in the absence of a point of care test, results will only become available after screening. Therefore these test results are not part of the eligibility criteria. However, they will be taken into account in analysing the results.

Ivermectin treatment strategy

Following recommendations 1 dose of 150 µg/kg Ivermectin (Mectizan®) will be administered orally, treatment will be directly observed (DOT). Ivermectin is generally well tolerated. Common side effects of ivermectin include fever, itching, skin rash, oedema, myalgia and head ache.

Anti-epileptic drug treatment strategy

Both treatment arms will receive anti-epileptic treatment according to a standardized protocol. Treatment will start with phenobarbital 100 mg once a day which may be increased to 150-200 mg per day after 2 months if there is insufficient seizure reduction (less than 50% reduction of seizure frequency). If there are contraindications for use of phenobarbital (intellectual or behavioural disorders) or persistent side effects, carbamazepine will be prescribed (in adults initial dose 100-200 mg per day, maintenance dose 400-1400 mg, in children initial dose is 5 mg/kg/day, maintenance dose 10-30 mg/kg day). In the case of side effects related to carbamazepine we will start with sodium valproate (in adults initial dose 400 mg/day, maintenance dose 400-2000 mg/day, in children initial dose 15-20 mg/kg/day and maintenance dose 15-30 mg/kg/day). In the case of carbamazepine and sodium valproate we will prescribe initial dose in all patients and will increase this to the lowest maintenance dose at 2 weeks visit. In case of dose-determined side effects dose reduction is permitted. Dose may be increased at the 2 months visit if there is insufficient seizure control (less than 50% reduction in seizure frequency). Individual treatment decisions will be made by the team physician who has received specific training in epilepsy treatment and can consult with the team neurologist. Patient and family will be informed on the following regarding epilepsy treatment;

* the delay in onset of effect and the time course of treatment;
* potential side-effects and the risk of these symptoms; to seek help promptly if these are distressing;
* the risk of abrupt discontinuation/withdrawal symptoms on missing doses;
* the need for regular follow-up.

Compliance

Indirect (pill count) and direct (AED blood levels) methods will be used to check for compliance to AED treatment. Community volunteers will be trained to assist the research team and local health team with the follow up of the trial participants and for compliance monitoring at the home of the participants. The centre visit at week 2 is scheduled to check for side effects in order to minimize withdrawal from AED treatment. Although non-compliant patients are expected to be equally distributed among treatment arms because of randomization, and therefore not to influence outcome, it is of importance to put effort in minimizing non-compliance. Community volunteers will also be trained to become community directed distributors of Ivermectin after completion of the trial.

Endpoints

Primary endpoint is proportion of patients who have achieved seizure freedom after 4 months. Seizure freedom will be defined as no seizures the last month of the trial (month 4). Secondary endpoints are proportion of patients at month 4 with >50 % reduction in seizure frequency compared to reported seizure frequency at randomization, and microfilarial load measured in skin snip. The seizure frequency data will be collected starting from day 1 using a "seizure diary". Reduction of seizures will be compared between Ivermectin and non-Ivermectin arms.

Baseline and follow-up procedures

At baseline information will be collected on seizure semiology, frequency, risk factors, treatment history and Ivermectin treatment in the past. A full physical and neurological examination will be performed together with serological testing and skin snip examination. Weight and height measurements will be carried out and the participants body mass index will be calculated at baseline and follow-up visits.Trial participants will be instructed how to fill out a seizure calendar and record intake of AEDs. Two weeks after randomization a centre visit is scheduled to assess potential side effects of AED. Side effects will be recorded using a structured questionnaire inquiring about known side effects of phenobarbital, carbamazepine or sodium valproate. To assess seizure frequency centre visits are scheduled after 2 weeks, 1, 2, 3 and 4 months. To minimize loss to follow-up we use GPS coordinates to locate study participants. During these visits neurological and physical examination will be repeated, adverse events will be evaluated and we will count AED pills for indirect measurement of AED compliance. At the 4th visit skin snip examination and OV serology will be repeated. Additionally, AED blood levels will be measured to directly assess AED compliance.

If a participant is not able to visit the study centre, a home visit will be performed to monitor AED use and seizure frequency.

Data Analysis

Sample size calculation

It is expected that 4 months of treatment with AEDs (phenobarbital, carbamazepine or sodium valproate) will lead to seizure freedom in 50 % of the patients (experience of R Idro in Uganda). In a clinical trial performed in Rethy (Ituri) comparing the safety and parasitological efficacy of Moxidectin vs Ivermectin treatment in persons with OV infection not receiving anti-epileptic treatment, 6 (80%) of 7 trial participants with epilepsy were seizure free at 4 months.

Null hypothesis: The probability of seizure freedom at 4 months for immediate Ivermectin treatment is equal to the probability of seizure freedom at months for delayed Ivermectin treatment. If we expect that seizure freedom at 4 months will be obtained in 50% of the participants with phenobarbital alone and that with additional Ivermectin treatment 80% of patients will achieve seizure freedom at 4 months, about 104 subjects (52 per group) are needed to achieve the power of 90% to reject the null hypothesis at the 5% significance level. Considering that 5% of the patients will be lost to follow up 110 patients will be enrolled in the trial.

All comparative analyses will be based on the intention- to- treat principle: all randomized patients will be included in the analysis according to the result of the randomization.

For the primary endpoint, the null hypothesis will be tested by comparing the observed proportion of responses in arm A with the corresponding proportion in arm B at the one sided 5% significance level by using the Cochran Mantel Haenszel test for comparison of two independent proportions. The Cochran Mantel Haenszel test will be performed controlling for baseline frequency of seizures. The same test will be used for the secondary end point. Change vs baseline in skin micofilarial load at month 4 will be analyzed by means of the T-test. Frequencies of seizures will be compared between participants with and without positive microfilaria skin snips at month 4.

Patients lost to follow up will be regarded as non-responders. Similarly, patients for whom the AED regimen had to be adapted because of an increasing number of seizures will be considered as non-responders. AED treatment changes because of side effects or possible interactions with other drugs will not be considered a treatment failure.

Data handling and record keeping

All relevant clinical information will be collected on tablets. The identity and information of trial participants is kept confidential. Data will be entered in a web-based electronic database, compliant with GCP, as defined by the International Conference on Harmonisation (ICH), that is access-controlled and data anonymized.

Monitoring, Oversight, and Reporting

The trial Sponsor is the University of Antwerp. The study team will undergo Good Clinical and Laboratory Practice (GCP, GCLP) training) protocol training and training in special procedures. An independent experienced clinical trial monitor will monitor the trial and report to the Sponsor. The monitoring will include checking the consent procedure, clinical event reporting, compliance with protocol SOPs, and treatment adherence. Data queries will be handled according to a quality management plan. A Data Safety Monitoring Board will be established to review safety, not for efficacy as early-stopping for efficacy is not considered. All adverse study drug reactions, serious adverse events and deaths will be reported to the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Age 5 years and above
* Signed informed consent form
* Normal neurological development until onset of epilepsy
* Onset of epilepsy between ages of 5 and 18 years
* Seizure frequency of ≥2 seizures per month
* Presence of microfilaria in skin snip and/or antibodies against Ov16

Exclusion Criteria:

* Ivermectin intake the last 9 months
* Pregnancy or breastfeeding
* Known or suspected allergy to Ivermectin
* Loa Loa microfilariae in blood
* Epilepsy with known cause (e.g. severe head trauma, perinatal asphyxia, patients with a history of cerebral malaria, meningitis or encephalitis)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
seizure freedom | 4 months
  absence of seizures month 4

SECONDARY OUTCOMES:
>50 % reduction in seizure frequency | 4 months
  >50 % reduction in seizure frequency compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Michel Mandro, MD, Principal Investigator — Chef de Bureau Inspection&Contrôle et Associé de Recherche Clinique
Locations (1):
- Centre de Recherche en Maladies Tropicales de l'Ituri, Rethy, Ituri, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
will be available at an ERC website
Supporting Information: Study Protocol, ICF
Time Frame: 10.01.19

REFERENCES:
- [Derived] Mandro M, Siewe Fodjo JN, Mukendi D, Dusabimana A, Menon S, Haesendonckx S, Lokonda R, Nakato S, Nyisi F, Abhafule G, Wonya'Rossi D, Jakwong JM, Suykerbuyk P, Meganck J, Hotterbeekx A, Colebunders R. Ivermectin as an adjuvant to anti-epileptic treatment in persons with onchocerciasis-associated epilepsy: A randomized proof-of-concept clinical trial. PLoS Negl Trop Dis. 2020 Jan 10;14(1):e0007966. doi: 10.1371/journal.pntd.0007966. eCollection 2020 Jan. PMID 31923177
- [Derived] Siewe Fodjo JN, Mandro M, Mukendi D, Tepage F, Menon S, Nakato S, Nyisi F, Abhafule G, Wonya'rossi D, Anyolito A, Lokonda R, Hotterbeekx A, Colebunders R. Onchocerciasis-associated epilepsy in the Democratic Republic of Congo: Clinical description and relationship with microfilarial density. PLoS Negl Trop Dis. 2019 Jul 17;13(7):e0007300. doi: 10.1371/journal.pntd.0007300. eCollection 2019 Jul. PMID 31314757
- [Derived] Colebunders R, Mandro M, Mukendi D, Dolo H, Suykerbuyk P, Van Oijen M. Ivermectin Treatment in Patients With Onchocerciasis-Associated Epilepsy: Protocol of a Randomized Clinical Trial. JMIR Res Protoc. 2017 Aug 30;6(8):e137. doi: 10.2196/resprot.7186. PMID 28855148